CLINICAL TRIAL: NCT01869920
Title: Effectiveness of an Educational Group Intervention in Primary Care to Maintain Exclusive Breastfeeding. Cluster Randomised Clinical Trial. PROLACT Study.
Brief Title: Effectiveness of an Educational Intervention to Maintain Exclusive Breastfeeding
Acronym: PROLACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Susana Martín Iglesias, Nurse, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI12/02609_PI12/02020
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Exclusive Breastfeeding
Keywords: breastfeeding; education; intervention
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): Intervention group receive a training education on breastfeeding. Education training is provided by an expert group from General Direction of Primary Care
  Interventions: Behavioral: Intervention group
- Controll group (Other): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Intervention group — Education on breastfeeding
  Arms: intervention group
Behavioral: Usual care — Usual care
  Arms: Controll group

SUMMARY:
Hypothesis: An educational intervention increases the proportion of mother-infant pairs using exclusive breastfeeding

DETAILED DESCRIPTION:
Objective: Evaluate the effectiveness of an educational group intervention performed by primary healthcare professionals in terms of increasing the proportion of mother-infant pairs using exclusive breastfeeding at six months compared to routine practice. Design: cluster randomized trial. Setting: Multicentre. Primary Care Health Centres (PCHC). Madrid. Subjects: mother-infant pairs using exclusive breastfeeding who come for any query to the health centre, as long as the infant is not older than four weeks and who consent to participate in the study.

Sample size: N= 432 (216 in each arm). Randomisation: Unit of randomization: primary healthcare centres.

Analysis unit: mother-infant pairs, recruitment to consecutive sampling. Intervention: Educational group intervention in the treatment group and the usual intervention in the control group.

Variables: Main response variable: mother-infant pairs using exclusive breastfeeding (EBF) at six months. Secondary variables: type of breastfeeding at 6 months, duration of EBF, reasons for ceasing breastfeeding, satisfaction with the intervention (SERVQUAL). Prognostic variables: infant, mother and professional.

Data Analysis: Analysis of main effectiveness by intention to treat, comparing the proportion of mother-infant pairs using EBF at six months in both groups. The estimation adjusted using an explanatory logistics regression model. To assess the effect of the educational group intervention on the duration of the various type of breastfeeding, a survival analysis will be used comparing the two groups using the log-rank test. The control of potential confounding variables will be performed by the construction of various Cox regression models.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years old or older,
* mother-infant pairs using exclusive breastfeeding,
* Signed Informed Consent

Exclusion Criteria:

* Any medical conditions that prevents breastfeeding
* infant should be not older than four weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding (EBF) | six months
  Evaluate the presence of EBF 6 months after educational intervention.

SECONDARY OUTCOMES:
Type of breastfeeding and duration of EBF | Six months
  EBF or not exclusive breastfeeding and duration in months
breastfeeding ceasing | During follow-up
  Reasons for breastfeeding ceasing

CONTACTS AND LOCATIONS:
Overall Officials: María J Santamaría, Nurse, Principal Investigator — Gerencia de Atención Primaria, Madrid; Susana Martín, Nurse, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia de Atencion Primaria, Madrid, Spain

REFERENCES:
- [Derived] Santamaria-Martin MJ, Martin-Iglesias S, Schwarz C, Rico-Blazquez M, Portocarrero-Nunez JA, Diez-Izquierdo L, Llamosas-Falcon L, Rodriguez-Barrientos R, Del-Cura-Gonzalez I; Grupo PROLACT. Effectiveness of a group educational intervention - prolact - in primary care to promote exclusive breastfeeding: a cluster randomized clinical trial. BMC Pregnancy Childbirth. 2022 Feb 16;22(1):132. doi: 10.1186/s12884-022-04394-8. PMID 35172775
- [Derived] Martin-Iglesias S, Santamaria-Martin MJ, Alonso-Alvarez A, Rico-Blazquez M, Del Cura-Gonzalez I, Rodriguez-Barrientosn R, Barbera-Martin A, Sanz-Cuesta T, Isabel Coghen-Vigueras M, de Antonio-Ramirez I, Durand-Rincon I, Garrido-Rodriguez F, Geijo-Rincon MJ, Mielgo-Salvador R, Morales-Montalva MS, Reviriego-Gutierrez MA, Rivero-Garrido C, Ruiz-Calabria M, Santamaria-Mechano MP, Santiago-Fernandez R, Sillero-Quintana MI, Soto-Almendro B, Terol-Claramonte M, Villa-Arranz M. Effectiveness of an educational group intervention in primary healthcare for continued exclusive breast-feeding: PROLACT study. BMC Pregnancy Childbirth. 2018 Feb 26;18(1):59. doi: 10.1186/s12884-018-1679-3. PMID 29482516